CLINICAL TRIAL: NCT00151073
Title: An Evaluation of Estramustine, Docetaxel and Zoledronate in Patients With Hormone-Refractory Adenocarcinoma of the Prostate
Brief Title: Estramustine, Docetaxel and Zoledronate Treatment in Hormone-Refractory Adenocarcinoma of the Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2001-051
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Hormone-Refractory Prostate Cancer
Keywords: Zometa; Prostate Cancer; Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid; Estramustine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoledronate Alone (Experimental): Zoledronate is given alone for the first cycle. All subsequent cycles consist of Docetaxel (70mg/m^2) given on day 2, Estramustine (280mg) given orally three times per day on days 1-3, and Zoledronate (4mg) given intravenously on day 2.
  Interventions: Drug: Zoledronic acid; Drug: Estramustine; Drug: Docetaxel
- Docetaxel and Estramustine (Experimental): Docetaxel and Estramustine are given for the first cycle of therapy. All subsequent cycles consist of Docetaxel (70mg/m^2) given on day 2, Estramustine (280mg) given orally three times per day on days 1-3, and Zoledronate (4mg) given intravenously on day 2.
  Interventions: Drug: Zoledronic acid; Drug: Estramustine; Drug: Docetaxel

INTERVENTIONS:
Drug: Zoledronic acid
  Other Names: Zometa; Zoledronate
Drug: Estramustine
Drug: Docetaxel

SUMMARY:
Purpose: The aim of this clinical trail is to evaluate the effectiveness of Zoledronate (Zometa) combined with Estramustine and Docetaxel (Taxotere) in the treatment of patients with hormone-refractory prostate cancer.

DETAILED DESCRIPTION:
Hormone refractory prostate cancer refers to advanced disease in which the patient no longer responds to conventional hormonal treatment. When hormone therapy is no longer successful, chemotherapy is a treatment option. However, current single-agent treatment has shown to have limited benefit. In this clinical trail, investigators are evaluating the effectiveness of Zoledronate(Zometa) combined with Estramustine and Docetaxel (Taxotere) in the treatment of patients with hormone refractory prostate cancer. Zometa is a bisphosphonate, and may reduce or delay skeletal complications caused by bone metastases. Estramustine and Taxotere are chemotherapy drugs that have shown activity in hormone refractory prostate cancer. Eligible patients will be randomized to receive Estramustine and Docetaxel (Taxotere) in combination with Zometa or Zometa given alone.

ELIGIBILITY:
All patients must have a histologic diagnosis of hormone-refractory adenocarcinoma of the prostate, and hormone refractory disease must be demonstrated by the appearance of new lesions on bone or CT scan and/or a rising PSA value. (No evidence of brain metastasis or untreated spinal cord compression.)

Patients on total androgen suppression therapy must undergo nonsteroidal antiandrogen withdrawal and demonstrate a rising PSA 4 weeks after withdrawal from flutamide and 6 weeks after withdrawal from bicalutamide.

Patient must not be undergoing current chemotherapy, biologic therapy, other investigational or alternative anti-cancer directed therapy or radiation therapy.

Prior radiation therapy must have completed more than 4 weeks prior to registration.

Patients may not have received prior taxane-based cytotoxic chemotherapy for hormone refractory disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2002-04; Primary Completion 2005-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The Percent Increase/Decrease in Bone Markers from Baseline to Cycle 2 Day 2 (Day 23) of Treatment | Cycle 2 Day 2 of Treatment (Day 23 of Treatment)
  To assess and compare the effect of zoledronate and docetaxel/estramustine on markers of bone metabolism in patients with hormone-refractory prostate cancer.

SECONDARY OUTCOMES:
Percentage of Patients that Respond to Treatment | Post 3 Cycles (63 days)
  A decrease in PSA of greater than or equal to 50%, without evidence of progression in the bones, will be considered as response to treatment.
The Number of Toxicities Experienced by Patients | 30 Days Post Treatment

CONTACTS AND LOCATIONS:
Overall Officials: David C. Smith, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States